CLINICAL TRIAL: NCT01604720
Title: Review: Analysis of the Sample Size Definitions in the Randomized Clinical Trials Included in Systematic Reviews of the Hepato-biliary Group of the Cochrane Collaboration
Brief Title: Sample Size Definition in Cochrane Hepato-Biliary Trials
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Lecco (Other)
Responsible Party: Principal Investigator, Agostino Colli, Head of Internal Medicine Department AO provincia di Lecco, Azienda Ospedaliera di Lecco
Other Study IDs: AOLecco002
Record Dates: First submitted 2012-05-14; First posted 2012-05-24 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Definition of Sample Size in Randomized Clinical Trial Assessing Liver Disease
Keywords: sample size; liver disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sample size definition provides important information, allowing the groundwork for transparent reporting. The sample predefinition allows the trial to be large enough to be able to address the question that is being asked.

The aim of the present study is to assess, in all the randomized controlled trials (RCT) included in the Cochrane Hepato-Biliary Group (CHBG) systematic reviews, the quality of reporting sample size the accuracy of the calculations, the accuracy of the a priori assumptions and the effect on the agreement with pooled results in meta-analyses.

DETAILED DESCRIPTION:
The investigators aim to answers to these questions

Questions

* How large a proportion of recent hepato-biliary RCTs does report an adequate sample size estimation?
* Primary outcome is clearly defined ? and clinical meaningful ?
* Is the sample size calculation based on the primary outcome ?
* Does the predicted control event rate coincide with the actual one?
* What is the predicted intervention effect?
* Are confidence intervals of primary outcome results reported? Is there evidence of difference between the two arms?
* Is the effect size so large (> 50%) to suggest post hoc definition ?
* What is the accepted error alpha and beta?
* How many study do not comply with the usual rule of alpha = 5% beta = 20%?
* Do trials with planned sample size do better than those without ? Is the overlap between CI results less frequent ? Are their results more frequently "statistical" significant ?
* Do trials with planned sample more frequently agree with pooled results in meta-analysis ?
* Has the protocol been published in a public register before inclusion of participant?
* How often is intention-to-treat analyses employed as primary analysis?
* How often is the trial results resting upon subgroup analysis?

Methods:

All the randomized clinical trials included in a systematic review of the Cochrane Hepato-biliary group (according to my search 272) were detected and retrieved. Only two arm, parallel group superiority randomised controlled trials with a single primary outcome.

The investigators excluded reports for which the study design was factorial, cluster, or crossover For all selected articles, the investigators systematically retrieved and assessed the full published report of the trial, any extra material or appendices available online, the study design article, if cited, and the details of online registration of the trial, if mentioned. A standardised data collection form was generated on the basis of a review of the literature and a priori discussion and tested by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Two arms, parallel group superiority randomised controlled trials with a single primary outcome,

Exclusion Criteria:

* Reports for which the study design was factorial, cluster, or crossover

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Randomized clinical trials included in systematic reviews of the hepato-biliary Group of the Cochrane Collaboration
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
proportion of reported sample size definitions | up to three months after retrievement and inclusion of all studies
  number of included studies with explicit sample size definition/ number of included studies

CONTACTS AND LOCATIONS:
Overall Officials: agostino colli, MD, Principal Investigator — AO provincia di lecco
Locations (1):
- Medicine Department A.Manzoni Hospital, Lecco, Italy